CLINICAL TRIAL: NCT01519427
Title: A Phase II Trial of MAP Kinase Inhibition With AZD6244 Hydrogen Sulfate in Combination With MK-2206 (Akt Inhibitor) in Patients With BRAF V600-Mutant Advanced Melanoma Whose Disease Has Progressed on Prior Therapy With a Selective BRAF Inhibitor (i.e., Vemurafenib, Dabrafenib, LGX818)
Brief Title: Selumetinib and Akt Inhibitor MK2206 in Treating Patients With Stage III or Stage IV Melanoma Who Failed Prior Therapy With Vemurafenib or Dabrafenib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to slow accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00238; NCI-2012-00238 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000722048; VICCMEL1120 (Other: Vanderbilt-Ingram Cancer Center); 8867 (Other: CTEP); N01CM00100 (NIH); 16950 (Other: H. Lee Moffitt Cancer Center); NCT01510444 (obsolete NCT alias)
Record Dates: First submitted 2012-01-25; First posted 2012-01-27 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-01

CONDITIONS: Recurrent Melanoma; Stage IIIA Melanoma; Stage IIIB Melanoma; Stage IIIC Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — MK 2206; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (selumetinib and Akt inhibitor MK2206) (Experimental): Patients receive selumetinib PO BID on days 1-21 and Akt inhibitor MK2206 PO once weekly.
  Interventions: Drug: Akt inhibitor MK2206; Drug: selumetinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: Akt inhibitor MK2206 — Given PO
  Other Names: MK2206
Drug: selumetinib — Given PO
  Other Names: ARRY-142886; AZD6244
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well selumetinib and Akt inhibitor MK2206 works in treating patients with stage III or stage IV melanoma who failed prior therapy with vemurafenib or dabrafenib. Selumetinib and Akt inhibitor MK2206 stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet know whether giving selumetinib and Akt inhibitor MK2206 together is an effective treatment for advanced melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the frequency of objective clinical responses by RECIST 1.1 for these melanoma patients who have previously progressed on selective BRAF inhibitors when treated with MEK inhibitor, AZD6244 hydrogen sulfate plus Akt inhibitor, MK-2206.

II. To further characterize toxicities of both regimens in these patients who have progressed after BRAF inhibitor therapy.

SECONDARY OBJECTIVES:

I. With required fresh pretreatment biopsies on all patients, we plan to characterize the molecular state (genetic and proteomic) associated with BRAF inhibitor resistance. This may include an analysis of pathway activation, PI3/Akt or MAP kinase pathway; loss of expression of PTEN, secondary mutations in BRAF, other mutations in the MAP kinase pathway (NRAS, KRAS, HRAS, CRAF, MEK), activation of other RTKs (amplification, over expression, phosphorylation).

OUTLINE:

Patients receive selumetinib orally (PO) twice daily (BID) on days 1-21 and Akt inhibitor MK2206 PO once weekly.

After completion of study treatment, patients are followed up every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have incurable unresectable stage III or IV histologically confirmed Melanoma with V600-mutant BRAF disease and must have progressed after therapy on selective BRAF inhibitor; all patients must have biopsiable tumor and a biopsy must be performed with the collection of FFPE and if possible FF prior to initiation of treatment on this protocol; archival tumor tissue must also be obtained if at all available; this required biopsy will not be necessary if a previous biopsy of progressing tumor after selective BRAF therapy had already been obtained and is adequate
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral computed tomography (CT) scan
* Patients must have received prior therapy and progressed following a selective BRAF inhibitor (i.e., vemurafenib, dabrafenib, LGX818, etc.); patients must have completed prior therapy a minimum of 4 weeks previously (6 weeks for BCNU and/or mitomycin C), 4 weeks for prior biologic therapy, and 2 weeks for localized radiation therapy; all treatment related toxicity must have resolved to grade 2 or less as well; patients may initiate the protocol treatment at 48 hours following the completion of BRAF inhibitor; patients must have had no more than 2 prior chemotherapy regimens; patients cannot receive chemotherapy after the BRAF inhibitor treatment and prior to enrollment on this protocol; up to two prior immunotherapy regimens for advanced disease are allowed and one may be given between BRAF inhibitor therapy and this trial
* Patients must not be refractory to the BRAF inhibitor; patients must demonstrate some degree of tumor regression initially on BRAF inhibitor prior to progression; (tumor regression does not require RECIST objective response); they cannot have progressive disease at the time of first evaluation (4 or 8 weeks) on the BRAF inhibitor
* Baseline Ophthalmologic exam must be done at screening to include slit lamp exam and fundoscopy; an OCT scan should be considered in case of retinal abnormality at exam
* Life expectancy of greater than or equal to 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1 (Karnofsky ≥ 70%)
* Absolute neutrophil count ≥ 1,500 mm³
* Hemoglobin ≥ 9.0 g/dL (patients may be transfused to achieve level)
* Platelet count ≥ 100,000/μL
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvate transaminase(SGPT) < 2.5 X upper limit of normal (ULN)
* Total bilirubin < 1.5 mg/dL
* Serum creatinine ≤ 2.0 mg/dL OR creatinine clearance > 50 mL/min, determined by 24-hour urine collection
* Fasting blood glucose < 160 mg/dL OR
* HgbA1C < 8% disease (uncontrolled diabetes)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Patients must have a negative serum pregnancy test prior to being eligible to take part in the study
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with AZD6244 hydrogen sulfate and MK-2206
* Baseline echocardiogram or MUGA must be performed at screening and patients must have LVEF > 55%; additionally baseline EKG must be performed and corrected QTc must be < 480 milliseconds
* Baseline electrocardiogram(EKG) must be performed and corrected QTc must be < 480 milliseconds
* Patients must be able to swallow tablets and capsules to participate in the study
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD6244 hydrogen sulfate, MK-2206, or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, psychiatric illness/social situations that would limit compliance with study requirements, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension (BP >= 150/95 despite optimal therapy), baseline ejection fraction < 55% or the lower limit of institutional normal, heart failure NYHA Class II or above, prior or current cardiomyopathy, atrial fibrillation with heart rate > 100 bpm, and uncontrolled angina (Canadian Cardiovascular society grade II-IV despite medical therapy); acute coronary syndrome within 6 months from starting therapy
* Patients must have completed prior therapy a minimum of 4 weeks previously (6 weeks for BCNU and/or mitomycin C), 4 weeks for prior biologic therapy, and 2 weeks for localized radiation therapy
* All treatment-related toxicity must have resolved to grade 2 or less
* No patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients must have had no more than 2 prior chemotherapy regimens
* Patients cannot receive chemotherapy after the BRAF-inhibitor treatment and prior to enrollment on this protocol
* Up to two prior immunotherapy regimens for advanced disease are allowed and one may be given between BRAF-inhibitor therapy and this trial
* Patients may not be receiving any other investigational agents at the same time as study treatment
* Patients receiving medications or substances that are strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) are ineligible
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients must not have received chemotherapy in the time between the failure of BRAF inhibitor and the enrollment onto the present trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Sosman, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from January 2012 through February 2013.
Pre-assignment Details: Four potential subjects consented. Two were ineligible.
Period: Overall Study
Arm/Group | Treatment (Selumetinib and Akt Inhibitor MK2206)
Started | 2
Completed | 0
Not Completed | 2
Not completed — disease progression | 2

BASELINE CHARACTERISTICS:
Population: 2 consented patients were not eligible for the trial
Arm/Group | Treatment (Selumetinib and Akt Inhibitor MK2206)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response
Description: Number of patients in each response category, per Response Evaluation in Solid Tumors (RECIST) v.1.1: complete response (CR), disappearance of target lesions; partial response (PR) >=30% decrease in sum of longest diameter (LD) of target lesions; progressive disease (PD), >=20% increase in sum of LD of target lesions or appearance of new lesions; stable disease (SD), insufficient change in target lesions or new lesions to qualify as either PD or PR. Patients are categorized according to the best response achieved prior to occurrence of progressive disease, where best response hierarchy is CR>PR>SD>PD.
Time Frame: On-treatment date to date of progressive disease (assessed up to 30 days after end of treatment)
Population: All patients with best overall response data; patients are excluded if best overall response data is missing or if the patient is non-evaluable for best overall response.
Measure: Number; unit: participants
Arm/Group | Treatment (Selumetinib and Akt Inhibitor MK2206)
Number analyzed (Participants) | 2
participants
  Complete response | 0
  Partial response | 0
  Progressive disease | 1
  Stable disease | 1

2. Secondary Outcome: Changes in Biomarker Expression
Description: Pre-treatment tumor biopsy tissue and blood and day 7-14 tumor biopsy tissue and blood will be examined by immunohistochemistry for expression and phosphorylation of the proteins pERK, pMEK, pAKT, Ki67, pRpS6, CRAF, cyclin D, PDGFr, pPDGFr. IGFr1, and COT/Tp12 for changes from baseline
Time Frame: Before initiation of treatment and at 7-14 days, up to 2 years
Population: This clinical trial was terminated early. The investigators did not perform any biomarker expression analyses.
Arm/Group | Treatment (Selumetinib and Akt Inhibitor MK2206)
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Estimated probable duration of life without disease progression, from on-study date to earlier of progression date, or date of death from any cause, using the Kaplan-Meier method with censoring (see Analysis Population Description for additional details). Disease progression is defined by Response Evaluation in Solid Tumors (RECIST) v.1.1: >= 20% increase in sum of the longest diameter of target lesions, unequivocal progression of non-target lesions, or appearance of new lesions
Time Frame: On-study to lesser of date of progression or date of death from any cause, up to 2 years
Population: All patients are included in the analysis on intention-to-treat basis. Analysis is by Kaplan-Meier method, where either death or progression is an event, with censoring for non-progressed, non-expired patients at greater of off-study date or last known date alive.
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Selumetinib and Akt Inhibitor MK2206)
Number analyzed (Participants) | 2
days | 105 [42 to 168]

4. Secondary Outcome: Overall Survival
Description: Estimated probable duration of life from on-study date to date of death from any cause, using Kaplan-Meier method with censoring (see Analysis Population Description for additional details).
Time Frame: On-study date to date of death from any cause, up to 2 years
Population: All patients are included in the analysis on intention-to-treat basis. Analysis is by Kaplan-Meier method, where death is an event, with censoring for non-expired patients at greater of off-study date or last known alive date.
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Selumetinib and Akt Inhibitor MK2206)
Number analyzed (Participants) | 2
days | 153 [117 to 189]

ADVERSE EVENTS:
Time Frame: day 0 through day 168 (week 24)
Arm/Group | Treatment (Selumetinib and Akt Inhibitor MK2206)
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Selumetinib and Akt Inhibitor MK2206) (N=2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1)
pelvic pain (Musculoskeletal and connective tissue disorders) | 1 (1)
acute renal failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Selumetinib and Akt Inhibitor MK2206) (N=2)
lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (2)
anemia (Blood and lymphatic system disorders) | 1 (5)
electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
bladder infection (Infections and infestations) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1)
alanine aminotransferase increased (Investigations) | 2 (6)
aspartate aminotransferase increased (Investigations) | 1 (2)
creatinine increased (Investigations) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 2 (5)
hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3)
hypokalemia (Metabolism and nutrition disorders) | 1 (2)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
pain (General disorders) | 2 (2)
blurred vision (Eye disorders) | 1 (1)
pain eye (Eye disorders) | 1 (2)
hematuria (Renal and urinary disorders) | 1 (1)
rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
lymphedema (Vascular disorders) | 1 (1)
chills (General disorders) | 1 (1)
fatigue (General disorders) | 1 (2)
pain extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Because this study terminated early due to slow accrual, data were available for only the two eligible patients that enrolled before study closure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less